CLINICAL TRIAL: NCT00221026
Title: A Multicenter, Open-Label, Study of Extracorporeal Photoimmune Therapy With UVADEX in the Treatment of Patients With Moderately Active Crohn's Disease Who Are Refractory or Intolerant to Immunosuppressants and/or Anti-TNF Agents
Brief Title: Safety and Efficacy of Extracorporeal Photoimmune Therapy With UVADEX for the Treatment of Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD-2; NCT00105261 (obsolete NCT alias)
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Methoxsalen; Photopheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- drug (Experimental): ECP + Uvadex given for 12 weeks.
  Interventions: Drug: Methoxsalen +ECP; Procedure: Extracorporeal Photopheresis

INTERVENTIONS:
Drug: Methoxsalen +ECP — ECP + Uvadex given at weeks 1-12 weeks.
  Other Names: Uvadex
Procedure: Extracorporeal Photopheresis — ECP given at weeks 1 through 12.
  Other Names: uvadex+ECP

SUMMARY:
his study will explore the safety and activity of ECP treatment with UVADEX in inducing a clinical response (i.e., a CDAI decrease greater than or equal to 100 from baseline and/or a CDAI < 150) over a 12-week period in moderately active Crohn's disease (CDAI greater than or equal to 220 to < 450) patients who are refractory or intolerant to immunosuppressants and/or anti-TNF agents. This study will also assess response to continued treatment during a 12-week Extension Period in patients who have a clinical response at Week 12 of the Treatment Period and elect to participate in the Extension Period.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent must be obtained prior to conducting any study procedure.
* Patients must be greater than or equal to 18 years of age.
* Patients must have a body weight greater than or equal to 40 kg (88 lb).
* Patients must have had Crohn's disease for at least 6 months duration (with colitis, ileitis, or ileocolitis) confirmed by radiography or endoscopy.
* Patients must have a CDAI greater than or equal to 220 to < 450.
* Patients must have a CRP concentration > 10.0 mg/L (1.0 mg/dL) or evidence of active inflammatory luminal Crohn's disease as demonstrated by superficial and/or deep ulcerations, pseudopolyps, and/or ulcerated stenosis on colonoscopy within 8 weeks of screening.
* Patients who are receiving corticosteroids must be on a prednisone equivalent dose less than or equal to 25 mg/day or an oral (PO) budesonide dose less than or equal to 9 mg/day.
* Patients who are receiving any of the following concomitant Crohn's disease medications must have been on a stable dose of these medications for the specified period of time PRIOR TO confirmation of eligibility (this time period may include screening): aminosalicylates, antibiotics, and immunosuppressants (i.e., 6 MP, MTX, or AZA) for at least 4 weeks; corticosteroids or PO budesonide for at least 2 weeks; anti-TNF agents (i.e., infliximab or adalimumab) for at least 8 weeks.
* Patients who have failed treatment with immunosuppressants and/or anti-TNF agents.
* Patients who have fistulae are permitted, provided: patients have predominantly luminal Crohn's disease, and fistulae are not associated with abscess formation.
* Patients must have a platelet count greater than or equal to 50,000/microL (50.0 x 109/L).
* Female patients must be: postmenopausal, surgically incapable of bearing children, or practicing an acceptable method of birth control (acceptable methods include hormonal contraceptives, intrauterine device, and spermicide and barrier). Abstinence or partner/spouse sterility may also qualify at the Investigator's discretion. If a female patient is of childbearing potential, she must have a negative urine pregnancy test at screening. Male patients must also commit to using adequate contraceptive precautions (condoms). All patients (both males and females of childbearing potential) must commit to using adequate contraceptive precautions throughout their participation in the study and for at least 3 months following their last ECP treatment
* Patients must be able and willing to comply with all study procedures.

Exclusion Criteria:

* Patients who are concomitantly using biologic agents other than anti-TNF agents; cyclosporine (CSA), tacrolimus (FK506), mycophenolate mofetil (MMF), or investigational Crohn's disease therapies.
* Patients who, in the opinion of the Investigator, may not be able to remain on a stable dose of a concomitant Crohn's disease medication during the 12-week Treatment Period.
* Patients with currently symptomatic untreated diarrhea, due to conditions other than inflammatory Crohn's disease (e.g., bacterial or parasitic gastroenteritis, bile salt diarrhea, or bacterial overgrowth).
* Patients with symptomatic intestinal strictures.
* Patients with stomas.
* Patients with other local manifestations of Crohn's disease such as abscesses, or other disease manifestations for which surgery might be indicated, or which might preclude utilization of a CDAI to assess response to therapy (such as "short gut" syndrome).
* Patients who are unable to tolerate the extracorporeal volume shifts associated with ECP treatment due to the presence of any of the following conditions: uncompensated congestive heart failure, pulmonary edema, severe chronic obstructive pulmonary disease, severe asthma, renal failure, or hepatic failure.
* Patients receiving total parenteral nutrition, as the sole source of nutrition, within 3 weeks of screening.
* Female patients whose hemoglobin (Hgb) is < 8.5 g/dL or male patients whose Hgb is < 10.0 g/dL at screening.
* Patients with a poor tolerability of venipuncture or a lack of adequate venous access for required treatments and blood sampling.
* Patients who have a known hypersensitivity or allergy to psoralen (methoxsalen).
* Patients who have a known hypersensitivity or allergy to both heparin and citrate products.
* Female patients who are pregnant and/or lactating.
* Patients who have been enrolled in any investigational study for the treatment of Crohn's disease within 4 weeks of enrollment for non biologic therapies and within 8 weeks of enrollment for biologic therapies.
* Patients who have any of the following: a co-existing melanoma, squamous cell skin carcinoma, aphakia, photosensitive disease (e.g., porphyria, systemic lupus erythematosus, or albinism), a white blood cell count > 25,000 mm3, a previous splenectomy, or a clinically significant coagulation disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2004-12; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Crohns Disease Activity Index | 12 weeks
  The CDAI is a questionaire giving the change of disease acitvity.This study wil llook or a decrease in CDAI score of at least 100.

CONTACTS AND LOCATIONS:
Locations (15):
- United States (4):
  - NIH, Bethesda, Maryland
  - Metropolitian Gastroenterology Group, Chevy Chase, Maryland
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Mount Sinai Medical Center, New York, New York
- General Hospital of Vienna, Vienna, Austria
- Belgium (2):
  - Hospital Erasme/ULB, Brussels
  - UZ Leuven, Leuven
- Germany (8):
  - Universitat St Josef, Bochum
  - Krankenhaus Duren gem.GmbH, Düren
  - Universitatsklinik Essen, Essen
  - Universitatsklinikum, Jena
  - Universitatsklinikum Mannheim, Mannheim
  - University Hospital Munich-Grosshadem, Munich
  - Klinikum Oldenberg, Oldenburg
  - Medizinische Universitatsklinik Ulm, Ulm